CLINICAL TRIAL: NCT03226665
Title: Ultrasound Emergency Diagnosis of Small Bowel Obstruction. An Observational Study
Brief Title: Ultrasound Emergency Diagnosis of Small Bowel Obstruction
Acronym: USBOW
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera, Universitaria Policlinico Vittorio Emanuele (Other)
Responsible Party: Principal Investigator, Guglielmo Trovato, MD, PhD, Professor of Medicine - Research Project Planning Unit, Azienda Ospedaliera, Universitaria Policlinico Vittorio Emanuele
Other Study IDs: USBOW
Record Dates: First submitted 2017-07-14; First posted 2017-07-24 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Obstruction Bowel
Keywords: obstruction; small bowel; ultrasound
MeSH Terms: conditions — Intestinal Obstruction; Bites and Stings | interventions — Ultrasonography; Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ultrasound — definition of prevalence of US detected obstruction in patients referred to an emergency facilities with symptoms potentially suggestive for such diagnosis.
  Moreover, which clue, if any, could reinforce the need of US intestinal study, such as anaemia, CRP, NLR, hypotension.
  This information is not yet available elsewhere. Moreover, in this context, sensitivity and specificity of ultrasound vs. confirm by CT and other procedures will make more sense and will be consequently assessed.
  Other Names: plain x-rays; computerized tomography

SUMMARY:
Small bowel obstruction (SBO) is a common presentation to the emergency department (ED) and represents 15% of hospital admissions for acute abdominal complaints.

Plain radiography, although traditionally recommended as the initial diagnostic imaging modality of choice, has a sensitivity of only 59% to 77%. When clinical and radiographic assessment is indeterminate, computed tomography (CT) becomes the test of choice due to its superior resolution and increased ability to identify both obstruction and its aetiology Aim: this is a prospective study in a sample of patients presenting to the emergency department (ED) with abdominal pain, vomiting, or other symptoms suggestive of a SBO (history of previous surgeries, constipation, abnormal bowel sounds, and abdominal distention). Patients will be evaluated with US prior to x-ray and CT, with possible diagnostic confirms by endoscopy or surgery.

DETAILED DESCRIPTION:
Primary outcome:

Our objective was to study the accuracy of emergency medicine bedside ultrasonography and in patients with suspected small bowel obstruction (SBO).

Secondary outcome:

assess the usefulness of the history and physical examination in the prediction of diagnosis

US Diagnostic criteria:

* Bowel lumen diameter >2.5cm
* Wall thickness > 4 mm
* Decreased/absent peristalsis
* Back/forth stool movements
* Free fluid

Methods The study is based on the assessment of all consecutive patients (19-75 years) presenting in the emergency department of Policlinico VE of the University of Catania (or to other affiliated Hospitals, such as Cannizzaro and/or Ragusa hospitals), which show clinical clues of small bowel obstruction (SBO). The criterion of enrolment is the casual referral to few previously identified physicians, skilled in TUS procedures and which accepted to take part to this study.

The most similar study on this topic demonstrates an extremely high accuracy of US in the diagnosis of intestinal obstruction, so that no actual power analysis can be done. The rationale of the present prospective study is the definition of prevalence of US detected obstruction in patients referred to an emergency facilities with symptoms potentially suggestive for such diagnosis.

Moreover, which clue, if any, such as anaemia, CRP, NLR, hypotension, could reinforce the need of US intestinal study.

This information is not yet available elsewhere. Moreover, in this context, sensitivity and specificity of ultrasound vs. confirm by CT and other procedures will make more sense and will be consequently assessed.

The secondary reason of this investigation is the attempt to detect which are the prevalence and the feature of under-diagnosis or over-diagnosis by US vs. the actual condition.

IMPLEMENTATION. This is a medium-term pilot study, non-interventional, which can be performed better as a single centre investigation, with few skilled and committed emergency physicians, than as a multicentre study, which would have the possible bias of relying on a mosaic or on scarcely skilled or motivated MDs.

ELIGIBILITY:
Inclusion Criteria:

* acute abdominal pain
* clinical clues of small bowel obstruction (SBO) according to symptoms and physical examination in the clinic

Exclusion Criteria:

* pregnancy
* post-surgical patients
* Trauma

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to the emergency facility with the clinical suspicion - before any imaging procedure - of small bowel obstruction
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Moreover, which clue, if any, such as anaemia, CRP, NLR, hypotension, could reinforce the need of US intestinal study. | 12 months
  According to the emergency referral protocols, patients that are assessed at the triage phase as likely to have any abdominal acute disease, including bowel occlusion, are preliminary studied by laboratory concurrently with the record of vital signs (blood pressure, electrocardiogram, pulse oxymetry). These information will be available during the actual visit of the Abdominal ultrasound in emergency may show fluid effusion, hemorrhagic or not, liver and/or gallbladder disease, spleen disease - possible leakage -, vascular disease (such as aneurism), inflammatory disease (Appendicitis, diverticulitis, Crohn's disease), masses and nodes (tumors, parasitic, others) and bowel occlusion . Clues, (anaemia, increased C-Reactive Protein, electrolyte abnormalities, clinical symptoms, hypotension) may reinforce the opportunity of US intestinal study, according also to the concordance with the subsequent confirmatory procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Guglielmo Trovato, MD, Study Director — AOVE Policlininico unict

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guttman J, Stone MB, Kimberly HH, Rempell JS. Point-of-care ultrasonography for the diagnosis of small bowel obstruction in the emergency department. CJEM. 2015 Mar;17(2):206-9. doi: 10.2310/8000.2014.141382. PMID 25927264
- [Result] Taylor MR, Lalani N. Adult small bowel obstruction. Acad Emerg Med. 2013 Jun;20(6):528-44. doi: 10.1111/acem.12150. PMID 23758299
- [Result] Jang TB, Schindler D, Kaji AH. Bedside ultrasonography for the detection of small bowel obstruction in the emergency department. Emerg Med J. 2011 Aug;28(8):676-8. doi: 10.1136/emj.2010.095729. Epub 2010 Aug 22. PMID 20732861